CLINICAL TRIAL: NCT01342692
Title: Randomized Phase II Trial Seeking the Most Promising Drug Association With Azacitidine- in Higher Risk Myelodysplastic Syndromes
Brief Title: Best Promising Drug Association With Azacitidine in Higher Risk Myelodysplastic Syndromes
Acronym: AZA-PLUS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P081225
Record Dates: First submitted 2011-04-21; First posted 2011-04-27 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: MDS
MeSH Terms: interventions — Azacitidine; Valproic Acid; Lenalidomide; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Azacitidine alone (Active Comparator)
  Interventions: Drug: Azacitidine
- Azacitidine +Valproic acid (Experimental)
  Interventions: Drug: Azacitidine associated with Valproic acid
- Azacitidine +Lenalidomide (Experimental)
  Interventions: Drug: Azacitidine associated with Lenalidomide
- Azacitidine + Idarubicine (Experimental)
  Interventions: Drug: Azacitidine associated with Idarubicine

INTERVENTIONS:
Drug: Azacitidine — 6 cycles of Azacitidine 75 mg/m2 subcutaneously daily for 7 days, every 4 weeks The first course will be started on day 1 regardless of the blood count. Subsequent courses will be scheduled every 4 weeks
  Arms: Azacitidine alone
Drug: Azacitidine associated with Valproic acid — 6 cycles of Azacitidine 75 mg/m2 subcutaneously daily for 7 days, every 4 weeks Valproic Acid (Depakine-Chrono®) (VPA) will be administered concomitantly for a minimum of 6 cycles.
  - In patients aged 60 years or less: VPA (25 mg/kg twice a day i.e. 50 mg/kg/d) administered orally, daily for 7 days (days 1-7)
  - In patients older than 60 years: VPA (17.5 mg/kg twice a day i.e. 35 mg/Kg/d) administered orally daily for 7 days (days 1-7)
  Arms: Azacitidine +Valproic acid
Drug: Azacitidine associated with Lenalidomide — 6 cycles of Azacitidine 75 mg/m2 subcutaneously daily for 7 days, every 4 weeks Lenalidomide (Revlimid®) will be administered once daily orally as continuous schedule started on day 1 of Azacitidine.
  Patients will receive Lenalidomide 10 mg/d, during 14 days (D1 to D14)
  Arms: Azacitidine +Lenalidomide
Drug: Azacitidine associated with Idarubicine — Azacitidine (Vidaza®) will be administered similarly to group 1 exposed above. Idarubicin (Zavedos®) as the reconstituted solution, will be administered slowly by the intravenous route over 60 minutes at 10 mg/m²of body-surface area on day 8 of Azacitidine or day 10 if azacitidine was administered according to (5-2-2 regimen)
  Arms: Azacitidine + Idarubicine

SUMMARY:
In order to improve the overall survival benefit observed with AZA in higher risk MDS, its combination with other active drugs in MDS must be tested.

Among drugs that have demonstrated to be active as a single agent in MDS and have preclinical potential additive or synergistic activity with AZA are Histone deacetylase (HDAC) inhibitors including Valproic acid, Lenalidomide and idarubicin. Phase I studies have already been conducted or are being conducted combining those agents to demethylating agents, showing a low toxicity profile and significant responses in high risk MDS. In this phase II randomized trial, we want to identify the most promising combination of Azacitidine and another drug (among 3 drugs: Valproic acid, Lenalidomide and Idarubicin) in higher risk MDS, by comparison to Azacitidine alone. Of note, based on efficacy and toxicity, one or several combinations may be stopped, and others, previously tested in phase I trials, included after protocol amendment.

DETAILED DESCRIPTION:
The main objective of this phase II randomized trial is to identify, among 3 combinations of Azacitidine and another drug evaluated simultaneously, the most promising combination(s) for the treatment of higher risk MDS (IPSS Int-2 and High) compared to Azacitidine alone. The 3 tested drugs in combination with Azacitidine are: Valproic Acid, Lenalidomide and Idarubicin.

The aim of this trial is to identify, in a situation where several potentially interesting drugs tested in combination with AZA exist, the most promising combination(s) based on efficacy compared to azacitidine alone, based on a two-stage design that allows a formal efficacy comparison between the K=3 investigational treatment groups and the control group.

ELIGIBILITY:
Inclusion Criteria:

* age>=18 years
* Must be able to adhere to the study visit schedule and other protocol requirements
* Documented diagnosis of MDS, including AREB-t according to FAB classification or CMML (with WBC < 13,000/mm3) that meets IPSS criteria for intermediate-2 or high-risk.
* Patients should be willing to use adequate contraceptive methods during all the duration of the study

Exclusion Criteria:

1. Treatment with AZA or Decitabine in the previous 6 months
2. Previous treatment with any HDAC inhibitor (Sodium valproate, Vorinostat, depsipeptide ou NSC-630176, MS 275, LAQ-824, PXD-101, LBH589, MGCD0103, CRA024781, etc). If Sodium Valproate (Depakine®) was used for seizure, a wash-out period of at least 30 days is required and an appropriate treatment replacement should be performed.
3. Ongoing treatment with corticosteroids exceeding 30mg of prednisone per day. A wash out period of at least 7 days is required.
4. HIV infection
5. Creatinine > 1.5 ULN
6. Serum AST or ALT > 3.0 x upper limit of normal (ULN)
7. Serum total bilirubin > 1.5 mg/dl (except for unconjugated hyperbilirubinemia due to Gilbert's disease or secondary to MDS).
8. ≥ grade-2 neuropathy
9. Previous history of Acute myeloblastic leukemia (with marrow blasts>30%)
10. Previous history of allogeneic stem cell transplantation
11. Contra-indication to Anthracyclines: Myocardiopathy, uncontrolled infection, serious renal or hepatic impairment; associated with yellow fever vaccine
12. Known hypersensitivity to the active substance or to any of the excipients of Vidaza®, of valproate, of divalproate, of valpromide, of Lenalidomide, of thalidomide, of idarubicin and/or anthracyclines
13. Patients with a history of severe congestive heart failure, clinically unstable cardiac or pulmonary disease
14. All hepatitis or known personal or familial severe hepatitis, particularly due to drugs
15. Depression with suicidal tendency
16. Use of MILLEPERTUIS, mefloquine
17. No medical insurance in the French Health system
18. Prior history of malignancy other than MDS (except basal cell or squamous cell carcinoma or carcinoma in situ of the cervix or breast) unless the subject has been free of disease for ≥ 3 years.
19. Pregnant or lactating females
20. Eligibility for allogeneic stem cell transplantation
21. very altered general condition , with WHO performance status of 4, or life expectancy of less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2011-06 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Remission, complete, partial or medullary after 6 cycles | 6 months
  Achievement of remission, complete, partial or medullary, according to the IWG 2006 criteria39 (see section 10 below) after 6 cycles

SECONDARY OUTCOMES:
Stable disease with hematological improvement | 3 and 6 months
  Achievement of stable disease with hematological improvement (HI), according to IWG 2006 criteria after 3 and 6 cycles
Duration of response | within 3 years
  Duration of response
Progression to acute myeloid leukemia | 3 years
Overall survival | 3 years
Number of adverse events | 3 years
  Number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Fenaux, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Avicenne hospital, Bobigny, France

REFERENCES:
- [Derived] Jacob L, Uvarova M, Boulet S, Begaj I, Chevret S. Evaluation of a multi-arm multi-stage Bayesian design for phase II drug selection trials - an example in hemato-oncology. BMC Med Res Methodol. 2016 Jun 2;16:67. doi: 10.1186/s12874-016-0166-7. PMID 27250349